CLINICAL TRIAL: NCT07009054
Title: Program for the Promotion of Physical Exercise and Healthy Eating (PEFAS) Culturally and Linguistically Adapted to the Population of Pakistani Origin With Obesity
Brief Title: Program for the Promotion of Physical Exercise and Healthy Eating Among Population of Pakistani Origin With Obesity
Acronym: PEFAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: University of Vic - Central University of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEFAS
Record Dates: First submitted 2024-11-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: obesity; metabolic syndrome; diet
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Nutrition Assessment; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Life-style interventions (diet and exercise)
  Interventions: Behavioral: Nutrition Education and Exercise
- Control (Other): Usual care
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Nutrition Education and Exercise — A 6-week intensive randomized controlled trial will be conducted with a total of 60 participants. Thirty participants will be assigned to the intervention group and thirty to the control group through simple randomization using a table of random numbers. The intervention group will receive one weekly theoretical-practical nutrition education session in Urdu and one physical activity session based on Nordic walking per week, for a total of six nutrition sessions and six physical activity sessions over the 6-week period.
  Arms: Active
Behavioral: Usual Care Group — The control group will participate in 2 theoretical sessions of nutrition education and 2 of physical exercise.
  Other Names: Usual care
  Arms: Control

SUMMARY:
This randomized control trial aims to evaluate the effectiveness of a culturally and linguistically adapted nutrition education and physical exercise program on lifestyle (diet and exercise), metabolic parameters, and fat content and distribution of people of Pakistani origin with obesity residing in the North Metropolitan health area of Barcelona. The betterment of the mentioned parameters is expected to be greater in individuals from the intervention group who will receive a total of 12 sessions of nutrition education and physical exercise compared to the control group who will participate in only 4 sessions.

DETAILED DESCRIPTION:
This study aims to assess the impact of a culturally and linguistically adapted nutrition education and physical exercise program on the acquisition of heart-healthy habits (diet and exercise), various metabolic parameters (including glycemic and lipid markers), and the content and distribution of ectopic fat in individuals of Pakistani origin with obesity residing in the North Metropolitan Health Area of Barcelona.

A 6-week intensive randomized controlled trial (RCT) will be implemented with a total of 60 participants. Baseline data will be collected using both quantitative and qualitative methods by a multidisciplinary team of nutrition and nursing professionals. Quantitative methods will be employed to gather data on sociodemographic characteristics, health status, quality of life, clinical variables, body composition, eating habits, nutrition knowledge and skills, and physical activity. Qualitative methods will be used to adapt the intervention to the cultural and practical needs of participants and to explore variables such as eating habits and nutrition-related skills in greater depth.

Study data will be collected and managed using REDCap (Research Electronic Data Capture) tools hosted at Germans Trias i Pujol University Hospital.

Following baseline assessments, participants will be randomized into intervention (n=30) and control (n=30) groups using simple random assignment via a table of random numbers. The randomization sequence will be concealed in sealed, opaque envelopes labeled with participant codes.

The intervention group will receive one weekly theoretical-practical nutrition education session conducted in Urdu and one Nordic walking-based physical activity session per week, over a period of 6 weeks (totaling 6 nutrition sessions and 6 physical activity sessions). Nutrition education sessions will be conducted in the therapeutic kitchen of Germans Trias i Pujol University Hospital. Physical activity sessions will take place in public green spaces near participants' residential areas.

The control group will participate in two theoretical sessions of nutrition education and two sessions of physical activity.

After completion of the intervention (6 weeks), follow-up data collection will be conducted using the same quantitative and qualitative approaches applied at baseline. Follow-up assessments will also be repeated at 3 and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being of Pakistani origin
* Being Aged over 18 years
* Having obesity, defined as BMI ≥ 27 Kg/m2
* Being attended at the Saint Roc or Gorg Primary Care Centers, Endocrinology and Nutrition External Consultations at the Germans Trias i Pujol University Hospital (HUGTiP) or at the Specialized Care Center (Dr. Barraquer in St. Adrià and Dr. Robert in Badalona)
* Voluntarily accepting participation in the study.

Exclusion Criteria:

* Presenting a physical or mental illness that could prevent participation in the study.
* Presenting any pathology that could limit life expectancy in the short term.
* Pregnancy.
* Having a close family member included in the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Fat mass and total body mass measured by bioimpedance analysis | Baseline, 3 months and 6 months
  Body fat mass and total body mass will be quantified using bioimpedanciometry
Thickness of superficial and pre-peritoneal fat (mm) measured by ultrasound of the rectus abdominis | Baseline, 3 months, and 6 months
  Subcutaneous and pre-peritoneal fat thickness will be assessed using ultrasound imaging of the rectus abdominis muscle.
Quadriceps muscle thickness (mm) measured by ultrasound | Baseline, 3 months, and 6 months
  Muscle mass will be evaluated through ultrasound measurements of the quadriceps muscl
Body Mass Index (BMI) in kg/m² | Baseline, 3 months, and 6 months
  BMI will be calculated as weight in kilograms divided by height in meters squared (BMI = kg/m²). Weight will be measured using a calibrated digital scale, and height will be measured with a portable stadiometer.
Waist circumference (cm) | Baseline, 3 months, and 6 months
  Waist circumference will be measured at the midpoint between the lowest rib and the iliac crest using non-stretchable tape, recorded to the nearest 0.1 cm with the participant standing.
Physical exercise | Baseline, 3 months and 6 months
  The information related to the physical exercise will be gathered through the validated Urdu version of the International Physical Activity Questionnaire (IPAQ). Results will be reported as a continuous variable (MET minutes a week). Furthermore, participants from both the control and the intervention group will be provided with a smartwatch that will register their daily physical activity. The results will be presented in total minutes of intense and moderate physical activity per week.
Health-related quality of life | Baseline, 3 months and 6 months
  Perceived physical and mental health will be assessed using the 12-Item Short Form Survey (SF-12). The SF-12 is a self-reported outcome measure of health-related quality of life, widely used in various ethnic groups. It consists of 12 questions that are scored in various ways. The total score range is 12-47 (higher scores mean a worse outcome).
Fasting glucose level (mg/dL) | Baseline, 3 months, and 6 months
  Fasting glucose will be measured in serum samples using enzymatic methods.
Hemoglobin A1C (%) | Baseline, 3 months, and 6 months
  HbA1c will be measured from whole blood using high-performance liquid chromatography (HPLC).
Insulin (mIU/L) | Baseline, 3 months, and 6 months
  Fasting insulin concentration will be measured using electrochemiluminescence immunoassay.
Aspartate aminotransferase (AST)(UI/L) | Baseline, 3 months, 6 months
  AST will be measured via kinetic UV test using an automated analyzer.
Alanine aminotransferase (ALT)(UI/L) | Baseline, 3 months, 6 months
  ALT will be measured via kinetic UV test using an automated analyzer.
Gamma-glutamyl transferase (GGT)(UI/L) | Baseline, 3 months, 6 months
  GGT will be measured using enzymatic colorimetric methods.
Total cholesterol (mg/dL) | Baseline, 3 months, 6 months
  Total cholesterol will be measured using enzymatic colorimetric methods.
LDL cholesterol (mg/dL) | Baseline, 3 months, 6 months
  LDL-C will be measured directly via homogenous enzymatic assay.
HDL cholesterol (mg/dL) | Baseline, 3 months, 6 months
  HDL-C will be measured directly via homogenous enzymatic assay.
Adherence to Mediterranean Diet using modified MEDAS questionnaire | Baseline, 3 months, 6 months
  Adherence to the Mediterranean Diet will be assessed using a modified version of the 14-item Mediterranean Diet Adherence Screener (MEDAS), excluding the alcohol intake item (13 items total). Scores range from 0 to 13, with higher scores indicating better adherence. A score < 9 indicates low adherence; ≥ 9 indicates good adherence.. Unit of measure: score 0-13
Nutrient intake measured by 24-hour Dietary Recall | Baseline, 3 months, 6 months
  Nutrient and food group intake will be assessed using a structured 24-hour Dietary Recall (24HR), administered by trained staff. Data will be analyzed using nutritional analysis software to estimate daily intake. Unit of measure: grams, Kcal

SECONDARY OUTCOMES:
Sociodemographic data | Baseline
  A survey will be administered in which the following data will be collected:place of birth, reason for migration, years of residence in Catalonia, members of the family unit, type of academic studies, occupation, languages known and spoken, religion practiced, center of origin, previous participation in similar programs.
Clinical history | Baseline
  The following clinical data will be collected with the help of the medical history: age, sex, presence of arterial hypertension (year of diagnosis and treatment), dyslipidemia (year of diagnosis and treatment), cardiovascular disease (ischemic heart disease, cerebrovascular disease, peripheral arterial disease) (age at diagnosis), DM (year of diagnosis, usual treatment), microvascular complications (retinopathy, nephropathy, neuropathy).
Toxic habits | Baseline, 3 months and 6 months
  Through the survey smoking habits and alcohol intake (UBEs/week) will be recorded.
Nutrition knowledge | Baseline, 3 months and 6 months
  Dietary knowledge will be evaluated in an ad hoc questionnaire of 14 questions related to some dietary aspects that will have three possible answers: true, false and I don't know. The focus groups will also include questions related to the dietary knowledge of the participants.
Nutrition skills | Baseline, 3 months and 6 months
  Dietary skills will be evaluated based on an ad hoc questionnaire of 13 questions that will analyze the degree of difficulty they have faced in carrying out different actions related to aspects of nutrition (planning, purchasing, preparation, etc.) during the last 15 days. These questions could be answered as follows: no difficulty (1 point), little difficulty (2 points), some difficulty (3 points), quite a bit of difficulty (4 points), and a lot of difficulty (5 points), with a minimum value of 13 points and maximum of 65 points. Higher scores will indicate greater difficulty in performing dietary tasks.
Total sleep duration (minutes) | Baseline and 3 months
  Sleep duration will be objectively measured using a smartwatch device. Total minutes of sleep during the night will be recorded.
Sleep stages duration (minutes) | Baseline and 3 months
  Sleep stage data (light, deep, and REM sleep) will be recorded using a smartwatch, reporting the duration in minutes spent in each stage.
Sleep stages distribution (% of total sleep) | Baseline and 3 months
  The percentage of total sleep time spent in each sleep stage (light, deep, REM) will be calculated and reported.
Degree of hepatic steatosis measured by CAP (dB/m) | Baseline and 6 months
  Hepatic fat content will be assessed using the Controlled Attenuation Parameter (CAP) obtained via transient elastography (FibroScan®).
Liver stiffness measured by transient elastography (kPa) | Baseline and 6 months
  Liver fibrosis will be evaluated by measuring liver stiffness using transient elastography (FibroScan®).

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Teresa Julian, MD, Principal Investigator — Hospital Universitario Germans Trias i Pujol (Badalona)
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No